CLINICAL TRIAL: NCT03806959
Title: Interest of Pan Capsule (Small Bowel and Colon Video Capsule) in Symptomatic Patients Suspected of Irritable Bowel Syndrome Requiring Colonoscopy Phase A Feasibility
Brief Title: Interest of Pan Capsule in Symptomatic Patients Suspected of Irritable Bowel Syndrome Requiring Colonoscopy
Acronym: IPSILON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Avicenne (Other)
Collaborators: Adeprina (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Professor, MD, PhD, Hospital Avicenne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A03229-44
Record Dates: First submitted 2019-01-10; First posted 2019-01-16 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: every patient will have both pan-capsule and colonoscopy. comparison intra-group between lesions found by the two examinations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pan Capsule and colonoscopy (Experimental): Every patient will have both Pan Capsule and colonoscopy examinations Descriptive study only
  Interventions: Other: Pan Capsule and colonoscopy in patients with IBS

INTERVENTIONS:
Other: Pan Capsule and colonoscopy in patients with IBS — Every patient will have both Pan Capsule and colonoscopy examinations Descriptive study only Usual biological tests (CBC, CRP, TSH, anti-transglutaminase antibodies) and measurement of fecal calprotectin.

SUMMARY:
Irritable bowel syndrome (IBS) is a chronic disease characterized by the association of abdominal pain and transit disorders. IBS affects 5 to 10% of the population. There are several forms of IBS: IBS-D (with predominant diarrhea), IBS-C (with constipation predominant) and IBS-M (mixed with alternating diarrhea and constipation). In the absence of a diagnostic test to confirm the existence of this syndrome, the diagnosis of IBS is based on clinical criteria (Rome IV criteria). In patients suspected of IBS, especially in patients with diarrhea (IBS-D or IBS-M), a colonoscopy with biopsies is often proposed in addition to biological tests (Complete Blood Count, C-reactive protein, thyroid stimulating hormon and anti-transglutaminase antibodies) by the physician or gastroenterologist to exclude an organic digestive disease such as celiac disease, IBD (Crohn's disease or ulcerative colitis), microscopic colitis or even neoplasia.

The colonoscopy is an invasive exploration and does not allow exploration of the entire small bowel.

The development of capsules allowed the exploration of the small bowel more recently of the colon. The new developed pan-capsule allows evaluation of both small bowel and colon.

The aim of this work is to evaluate in patients younger than 50 years, presenting suspicious digestive symptoms of IBS with diarrhea, the interest of a strategy based on the pan-capsule as an alternative to colonoscopy to eliminate a diagnosis of organic digestive disease (celiac disease, IBD, neoplasia, ..).

ELIGIBILITY:
Inclusion Criteria:

* Male or female: Age ≥ 18 years and ≤ 50 years
* Patients with symptoms compatible with IBS-D or IBS-M according to the treating physician.
* Indication for colonoscopy according to the physician
* Absence of prior colonoscopy
* Patient affiliated to a social security Insurance
* Signature of signed informed consent.

Exclusion Criteria:

* Functional or organic disorders of swallowing.
* Dysphagia or suspicion of digestive stenosis.
* Known Zenker Diverticule.
* Major surgical history of the digestive tract (exclusion of appendectomy, cholecystectomy, surgery of hemorrhoids).
* Known illness that could explain digestive symptoms.
* Symptoms suggestive of occlusion.
* Alteration of the general state and / or dehydration.
* Chronic uncontrolled disease.
* Disorders of consciousness.
* Uncontrolled heart disease: myocardial infarction in the last 6 months, anginal disease status, NYHA grade III and above congestive heart failure, ventricular tachycardia, ventricular fibrillation, severe heart block.
* Patient with a pacemaker or other implantable electronic medical device.
* Polyethylene glycol allergy.
* Oral iron intake in the four days preceding the video capsule.
* Pregnant or lactating woman, woman of childbearing age who has not performed a pregnancy test, women and men of childbearing potential without effective contraception.
* Impossible follow up for psychological or geographical reasons.
* Patient under safeguard of justice.
* Patient under guardianship or curatorship.
* Simultaneous participation in another clinical study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with digestive pathology and / or significant gastrointestinal lesion. | 1 month
  Number of patients with digestive pathology and / or significant gastrointestinal lesion (mucosal atrophy, mucosal erythema or ulceration, inflammatory bowel disease, neoplasia: colon adenocarcinoma, polyps> 5 mm, microscopic colitis).

SECONDARY OUTCOMES:
Acceptability of the pan-capsule, preference of one of the carried out explorations (pan-capsule or iléo-colonoscopy). | 1 month
  Index of acceptability (visual analogy scale)
Acceptability to complete the questionnaires (number of completed questionnaires). | 1 month
  Number of completed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert BENAMOUZIG, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre de Recherche sur Volontaires (CRV), Hospital Avicenne, Bobigny, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Pluart D, Sabate JM, Bouchoucha M, Hercberg S, Benamouzig R, Julia C. Functional gastrointestinal disorders in 35,447 adults and their association with body mass index. Aliment Pharmacol Ther. 2015 Apr;41(8):758-67. doi: 10.1111/apt.13143. Epub 2015 Mar 1. PMID 25728697
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Gralnek IM, Hays RD, Kilbourne A, Naliboff B, Mayer EA. The impact of irritable bowel syndrome on health-related quality of life. Gastroenterology. 2000 Sep;119(3):654-60. doi: 10.1053/gast.2000.16484. PMID 10982758
- [Background] Canavan C, West J, Card T. Review article: the economic impact of the irritable bowel syndrome. Aliment Pharmacol Ther. 2014 Nov;40(9):1023-34. doi: 10.1111/apt.12938. Epub 2014 Sep 9. PMID 25199904
- [Background] Corsetti M, Van Oudenhove L, Tack J. The quest for biomarkers in IBS-where should it lead us? Neurogastroenterol Motil. 2014 Dec;26(12):1669-76. doi: 10.1111/nmo.12475. PMID 25424580
- [Background] Andresen V, Whorwell P, Fortea J, Auziere S. An exploration of the barriers to the confident diagnosis of irritable bowel syndrome: A survey among general practitioners, gastroenterologists and experts in five European countries. United European Gastroenterol J. 2015 Feb;3(1):39-52. doi: 10.1177/2050640614558344. PMID 25653858
- [Background] Quigley EM. Overlapping irritable bowel syndrome and inflammatory bowel disease: less to this than meets the eye? Therap Adv Gastroenterol. 2016 Mar;9(2):199-212. doi: 10.1177/1756283X15621230. PMID 26929782
- [Background] Spiller R, Camilleri M, Longstreth GF. Do the symptom-based, Rome criteria of irritable bowel syndrome lead to better diagnosis and treatment outcomes? Clin Gastroenterol Hepatol. 2010 Feb;8(2):125-9; discussion 129-36. doi: 10.1016/j.cgh.2009.12.018. No abstract available. PMID 20152787
- [Background] Lieberman DA, Holub J, Eisen G, Kraemer D, Morris CD. Utilization of colonoscopy in the United States: results from a national consortium. Gastrointest Endosc. 2005 Dec;62(6):875-83. doi: 10.1016/j.gie.2005.06.037. PMID 16301030
- [Background] Chey WD, Nojkov B, Rubenstein JH, Dobhan RR, Greenson JK, Cash BD. The yield of colonoscopy in patients with non-constipated irritable bowel syndrome: results from a prospective, controlled US trial. Am J Gastroenterol. 2010 Apr;105(4):859-65. doi: 10.1038/ajg.2010.55. Epub 2010 Feb 23. PMID 20179696
- [Background] Ishihara S, Yashima K, Kushiyama Y, Izumi A, Kawashima K, Fujishiro H, Kojo H, Komazawa Y, Hamamoto T, Yamamoto T, Sasaki Y, Shimizu T, Okamoto E, Yoshimura T, Furuta K, Noguchi N, Tanaka H, Murawaki Y, Kinoshita Y. Prevalence of organic colonic lesions in patients meeting Rome III criteria for diagnosis of IBS: a prospective multi-center study utilizing colonoscopy. J Gastroenterol. 2012 Oct;47(10):1084-90. doi: 10.1007/s00535-012-0573-4. Epub 2012 Mar 30. PMID 22460220
- [Background] Patel P, Bercik P, Morgan DG, Bolino C, Pintos-Sanchez MI, Moayyedi P, Ford AC. Prevalence of organic disease at colonoscopy in patients with symptoms compatible with irritable bowel syndrome: cross-sectional survey. Scand J Gastroenterol. 2015 Jul;50(7):816-23. doi: 10.3109/00365521.2015.1007079. Epub 2015 Jan 30. PMID 25636675
- [Background] Soubieres A, Wilson P, Poullis A, Wilkins J, Rance M. Burden of irritable bowel syndrome in an increasingly cost-aware National Health Service. Frontline Gastroenterol. 2015 Oct;6(4):246-251. doi: 10.1136/flgastro-2014-100542. Epub 2015 Feb 24. PMID 28839818
- [Background] Pimentel M, Purdy C, Magar R, Rezaie A. A Predictive Model to Estimate Cost Savings of a Novel Diagnostic Blood Panel for Diagnosis of Diarrhea-predominant Irritable Bowel Syndrome. Clin Ther. 2016 Jul;38(7):1638-1652.e9. doi: 10.1016/j.clinthera.2016.05.003. Epub 2016 May 31. PMID 27261204